CLINICAL TRIAL: NCT00005466
Title: Stroke and MI in Users of Estrogen/Progestogen
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4910; R01HL047043 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Cerebrovascular Accident; Myocardial Infarction; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Stroke; Myocardial Infarction

SUMMARY:
To estimate the relative risks of acute myocardial infarction (MI) and of stroke in postmenopausal users of estrogen/progestogen (E/P) combinations and to estimate the relative risks of MI and of stroke in users of estrogen alone.

DETAILED DESCRIPTION:
BACKGROUND:

Post-menopausal hormone use is becoming increasingly widespread based on evidence of the benefits of estrogen use for bone and the heart. However, because estrogen alone substantially increases the risk of endometrial cancer, estrogen users who have not undergone a hysterectomy are frequently also placed on a progestogen (E/P), a strategy that reduces the likelihood of endometrial cancer when compared with use of estrogen alone. In 1991, there were almost no data on the risk of cardiovascular disease in post-menopausal women who used E/P combinations.

DESIGN NARRATIVE:

The study had a case-control design, Cases were women hospitalized with MI or stroke in any of nine participating Northern California Kaiser Permanente hospitals in a 36 month period. For each case, one control, matched by year of birth, was selected at random from among members of the Kaiser Permanente Health Plan who were expected to use the same nine hospitals for their medical care. Information about use of estrogen, E/P combinations, past use of oral contraceptives, menopause, hysterectomy and oophorectomy, demographics, general health status, preventive health care, and cardiovascular risk factors were collected in interviews done of the subjects or, for fatal cases, a surrogate. Information about then current use of estrogen and E/P combinations were also gathered by reviewing medical records.

The investigators used conditional logistic regression analysis to estimate the relative risks of MI and of stroke in users of E/P combinations, taking into account prior oophorectomy and other potential confounders. They also estimated the risks of acute MI and of stroke in users of estrogen alone, accounting for prior oophorectomy and potential confounders.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-08; Study Completion 1995-07 (Actual)

REFERENCES:
- [Background] Petitti DB, Sidney S, Quesenberry CP Jr, Bernstein A. Ischemic stroke and use of estrogen and estrogen/progestogen as hormone replacement therapy. Stroke. 1998 Jan;29(1):23-8. doi: 10.1161/01.str.29.1.23. PMID 9445323
- [Background] Sidney S, Petitti DB, Quesenberry CP Jr. Myocardial infarction and the use of estrogen and estrogen-progestogen in postmenopausal women. Ann Intern Med. 1997 Oct 1;127(7):501-8. doi: 10.7326/0003-4819-127-7-199710010-00001. PMID 9313017